CLINICAL TRIAL: NCT06511479
Title: Telephone-based Mindfulness Training to Reduce Blood Pressure in Black Women With Hypertension in the Jackson Heart Study
Brief Title: Jackson Heart Study Women's Hypertension Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-00717; R01MD016402 (NIH)
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIND-BP (Experimental): Participants who are randomly assigned to receive the MIND-BP program, a virtually delivered mindfulness training group.
  Interventions: Behavioral: MIND-BP
- BOOST (Experimental): Participants who are randomly assigned to receive the BOOST program, a virtually delivered mindfulness training group.
  Interventions: Behavioral: BOOST

INTERVENTIONS:
Behavioral: MIND-BP — 8-week program delivered to small groups by a trained facilitator using Zoom/Webex. Each session is one hour long and includes a check-in period, teaching on the week's topic, group discussion, a skill-building exercise and home practice assignment. Participants receive a workbook of all session content, audio guides for home practice, and practice logs. At the start of the program, the stress response and its importance for hypertension and cardiovascular disease is discussed, and the rationale for the mindfulness and cognitive skills to be taught are explained. Weekly sessions focus on learning and practicing skills.
  Arms: MIND-BP
Behavioral: BOOST — The BOOST program is designed to control for attention, credibility, and expectation of benefit. To parallel MIND-BP, the BOOST program will be delivered in 8 weekly group sessions via Zoom/Webex and led by a trained facilitator. Each weekly BOOST session will be 1 hour long and comprised of a check-in period, introduction of the week's topic, and group discussion. Didactic information, skill-building instruction and home practice are not included. Weekly BOOST session topics include: (1) personal experience of hypertension; (2) personal experience of stress; (3) personal experience of mood-related challenges; (4) personal experience of social relationships; (5) concerns related to hypertension treatment; (6) concerns about other health problems; (7) personal experience related to healthcare; and (8) review of the BOOST experience.
  Arms: BOOST

SUMMARY:
High blood pressure is a powerful risk factor for heart disease. Black women are more likely to have high blood pressure than white women or Hispanic women. Even when they are aware they have high blood pressure, many people struggle to keep their blood pressure controlled. Research shows a connection between life stress and high blood pressure and heart disease outcomes. Mindfulness training programs can help people regulate their emotions and cope with stress. Research shows that mindfulness programs can also lower blood pressure. This study will compare two programs: MIND-BP, a Zoom-based mindfulness training group; and BOOST, a Zoom-based support group. The aims of the study are to test if the MIND-BP program leads to greater reductions in blood pressure, stress and depressive symptoms than the BOOST program in Black women with high blood pressure who are participating in the Jackson Heart Study. The primary outcome measure is 6-month change in systolic blood pressure. The secondary outcome measures are 6-month changes in perceived stress and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female participant in Jackson Heart Study
* Willing to be randomized and comply with all aspects of protocol
* Willing to be audio-recorded during group sessions.

Exclusion Criteria:

* Positive cognitive screen (MMSE <19)
* Severe depressive symptoms (CES-D ≥16)
* Pregnant or planning to become pregnant in the next 6 months
* Current participation in another trial
* Arm circumference >45 cm and <22 cm

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline, Month 6
  Change in average systolic blood pressure (SBP) from 7 consecutive days of home blood pressure monitoring.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) Score at Baseline | Baseline
  The 10-item Perceived Stress Scale (PSS-10) is a validated measure of perceived stress that assesses the degree to which situations in one's life are appraised as overwhelming, uncontrollable, and unpredictable over the last month. Items are rated on a 5-point scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 40; higher total scores indicate greater perceived stress.
Perceived Stress Scale (PSS-10) Score at Month 3 | Month 3
  The 10-item Perceived Stress Scale (PSS-10) is a validated measure of perceived stress that assesses the degree to which situations in one's life are appraised as overwhelming, uncontrollable, and unpredictable over the last month. Items are rated on a 5-point scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 40; higher total scores indicate greater perceived stress.
Perceived Stress Scale (PSS-10) Score at Month 6 | Month 6
  The 10-item Perceived Stress Scale (PSS-10) is a validated measure of perceived stress that assesses the degree to which situations in one's life are appraised as overwhelming, uncontrollable, and unpredictable over the last month. Items are rated on a 5-point scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 40; higher total scores indicate greater perceived stress.
Center for Epidemiological Studies Depression (CES-D) Score at Baseline | Baseline
  20-item assessment of the frequency of depressive symptoms during the prior week. Items are rated on a 4-point scale. The total score is the sum of responses and ranges from 0 to 60; higher total scores indicate greater frequency of depressive symptoms.
Center for Epidemiological Studies Depression (CES-D) Score at Month 3 | Month 3
  20-item assessment of the frequency of depressive symptoms during the prior week. Items are rated on a 4-point scale. The total score is the sum of responses and ranges from 0 to 60; higher total scores indicate greater frequency of depressive symptoms.
Center for Epidemiological Studies Depression (CES-D) Score at Month 6 | Month 6
  20-item assessment of the frequency of depressive symptoms during the prior week. Items are rated on a 4-point scale. The total score is the sum of responses and ranges from 0 to 60; higher total scores indicate greater frequency of depressive symptoms.
Number of Participants with Uncontrolled Hypertension at Baseline | Baseline
  Uncontrolled hypertension will be defined (using average blood pressure from 7 consecutive days of home blood pressure monitoring at each point) as mean SBP ≥130 mmHg or mean diastolic BP (DBP) ≥80 mmHg, as recommended in the 2017 American College of Cardiology/American Heart Association Guideline.
Number of Participants with Uncontrolled Hypertension at Month 3 | Month 3
  Uncontrolled hypertension will be defined (using average blood pressure from 7 consecutive days of home blood pressure monitoring at each point) as mean SBP ≥130 mmHg or mean diastolic BP (DBP) ≥80 mmHg, as recommended in the 2017 American College of Cardiology/American Heart Association Guideline.
Number of Participants with Uncontrolled Hypertension at Month 6 | Month 6
  Uncontrolled hypertension will be defined (using average blood pressure from 7 consecutive days of home blood pressure monitoring at each point) as mean SBP ≥130 mmHg or mean diastolic BP (DBP) ≥80 mmHg, as recommended in the 2017 American College of Cardiology/American Heart Association Guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared immediately following publication with no end date. The data will be shared with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose; the data are permitted to be used to achieve aims in the approved protocol. A data use agreement will be established between the investigator and the University of Mississippi Medical Center. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose will be permitted to access the data; the data are permitted to be used to achieve aims in the approved protocol. A data use agreement will be established between the investigator and the University of Mississippi Medical Center.